CLINICAL TRIAL: NCT05602922
Title: A Randomised Controlled Study of Liu-Zi-Jue Exercise Combined With Conventional Rehabilitation for Dysphagia in Post-stroke
Brief Title: Liu-Zi-Jue Exercise Combined With Conventional Rehabilitation Treat Dysphagia in Post-stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Ruijie Ma, Clinical Professor, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20220605105846789
Record Dates: First submitted 2022-09-25; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Stroke; Dysphagia
Keywords: stroke; dysphagia; rehabilitation; Liu-Zi-Jue Exercise
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- basic treatment+ swallowing rehabilitation treatment (Active Comparator): Swallowing function training mainly includes indirect training, direct training, and compensatory techniques, once a day for 20 minutes each time. In addition, a low-frequency electric VitalStim swallowing therapy device (produced by Chattanooga, USA) was also used for electrical stimulation therapy. The treatment parameters were 700ms in width, two-way square wave, 0～25mA in amplitude, and 30～80Hz in fixed frequency. The A electrode of channel 1 is placed above the hyoid bone, and the B electrode is placed above the notch on the thyroid cartilage. The channel 2 electrode C and electrode D of the therapeutic apparatus are arranged vertically and equidistantly according to the electrode A and electrode B. After the electrodes are placed, turn on the power. The stimulation intensity is based on the maximum stimulation that the patient can tolerate. 1 time a day, 30min each time, a total of 4 weeks.
  Interventions: Other: Basic treatment +Swallowing rehabilitation training
- basic treatment+ swallowing rehabilitation treatment+ Liu-Zi-Jue (Experimental): On the basis of the control group, the Liu-Zi-Jue exercises were performed, including "Xu, He, Hu, Si, Chui, Xi", 6 times each time, 5 times a week, each exercise for 30 minutes, and continuous treatment for 4 weeks.
  Interventions: Combination Product: Liu-Zi-Jue Exercise

INTERVENTIONS:
Combination Product: Liu-Zi-Jue Exercise — Combined with the actual situation of stroke patients, this Liu-Zi-Jue Exercise adopts the sitting position.
  Arms: basic treatment+ swallowing rehabilitation treatment+ Liu-Zi-Jue
Other: Basic treatment +Swallowing rehabilitation training — Basic treatment +Swallowing rehabilitation training
  Arms: basic treatment+ swallowing rehabilitation treatment

SUMMARY:
In this study, a prospective, randomized controlled method was adopted, with patients with post-stroke dysphagia as the main research objects, applying "Liu-Zi-Jue" to the patients for rehabilitation intervention, and to explore the effect of "Liu-Zi-Jue" on the swallowing function of patients with post-stroke dysphagia. In order to provide a safe and effective TCM treatment plan for patients with dysphagia after stroke, reduce the disability rate after stroke and improve the quality of life of patients.

DETAILED DESCRIPTION:
This study is a single-center, prospective, randomized, controlled, clinical trial. A total of 60 inpatients with post-stroke dysphagia in the Third Affiliated Hospital of Zhejiang Chinese Medical University from April 2022 to December 2023 will be selected, and the patients will be assigned to the experimental group and the control group with 30 cases in each group according to the random number table. The control group will be given basic treatment and swallowing rehabilitation therapy, while the experimental group will be given Liu-Zi-Jue Exercise on the basis of the control group. Both groups are going to treat for 4 weeks and follow up for 60 days. Standardized Swallowing Assessment, Video Fluoroscopic Swallowing Study, Volume Viscosity Swallow Test, Penetration-aspiration scale, Water Swallow Test, Modified Barthel Index will be used to evaluate the swallowing function and living ability of patients, and to evaluate the clinical effect of Liu-Zi-Jue Exercise training on patients with dysphagia after stroke. Efficacy, clear its treatment advantages, in order to optimize the cost-effective and standardized rehabilitation program for dysphagia during stroke recovery, improve patients' swallowing function, improve their activities of daily living, and minimize the waste of health resources.

ELIGIBILITY:
Inclusion Criteria:

1.Meeting the diagnostic criteria of stroke in traditional Chinese medicine. 2.Meeting the diagnostic criteria of ischemic stroke in Western medicine. 3.Meeting the diagnostic criteria for swallowing disorders. 4.30 ≤ age ≤ 85 years; gender not restricted. 5.Duration of illness ≤ 180 days. 6.Water test at level 3 and above. 7.Voluntary participation in the subject, no serious complications, acceptable and good compliance with Liu-Zi-Jue Exercise treatment.

8.Sign the informed consent form.

Exclusion Criteria:

1. Patients with true bulbar palsy caused by brainstem encephalitis, motor neuron disease, pontine extension tumor, multiple sclerosis, myasthenia gravis, syringomyelia, etc.
2. Cerebrovascular malformation, trauma, aneurysm, etc.
3. Pregnant or lactating women.
4. Patients with severe primary chronic diseases such as heart, liver, kidney and other organs, as well as endocrine system and hematopoietic system, severe dementia and cognitive impairment (Simple Mental State Scale Examination (MMSE): score <15 points), severe language comprehension disorder, mentally ill patients.
5. Patients with various bleeding tendency diseases.
6. Patients who are allergic to swallowing contrast drugs.
7. Patients who do not meet the inclusion criteria, do not have poor treatment compliance as prescribed, cannot judge the efficacy or have incomplete data, which affect the judgment of efficacy and are not suitable for clinical observation.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Change in Standardized Swallowing Assessment | Baseline, 4 weeks and 60 days
  The scale consists of 3 parts, the first part includes the overall evaluation of the patient's consciousness, lip closure control, head and trunk control, breathing pattern, soft palate movement, posterior function, gag reflex, spontaneous cough, etc., with a total of 8-23 points; Part 2: Let the patient drink 5ml of water, repeat 3 times, observe the water flow at the corners of the mouth when drinking water, laryngeal movement during swallowing, repeated swallowing, wheezing and laryngeal function, a total of 5 to 11 points; in the second part, if 2 or more times swallowing is normal Then carry out the third part of the assessment: the patient drinks 60 ml of water, and observes the drinking and swallowing, with a total of 5 to 12 points. The total score of this scale is 18-46 points, and the higher the score, the worse the swallowing function.

SECONDARY OUTCOMES:
Video fluoroscopic swallowing study | Baseline and 4 weeks
  The scale mainly includes three parts: oral stage, pharyngeal stage, and the degree of aspiration. The oral stage is 0-2 points; the pharyngeal stage is 0-3, and the degree of aspiration is 0-4. The total score is 9 points. The higher the value, the better the swallowing function.
The volume viscosity swallow test | Baseline and 4 weeks
  The volume selected during the test is a small amount (5ml), a medium amount (10ml), a large amount (20ml), and the consistency is low consistency (water sample), medium consistency (thick paste), high consistency (pudding), according to different Combination, the complete test requires a total of 9 mouthfuls to eat, observe whether the patient coughs, whether the sound quality changes, and whether the blood oxygen saturation decreases to determine the patient's swallowing safety, observe the patient's lip closure, oral cavity residue, pharyngeal residue, and divided swallowing to determine the patient's swallowing status Effectiveness to analyze the risk of swallowing and eating in patients.
Penetration-aspiration scale | Baseline and 4 weeks
  The scale is divided into 3 categories and 8 grades according to whether the contrast agent enters the airway, the depth of entering the airway, and whether it can be discharged.
Water swallow test | Before treatment, after 4 weeks of treatment and after 60 days of treatment.
  The patient sits, drinks 30 ml of warm water, and is divided into 5 grades according to the time required and the condition of choking.
Modified Barthel Index | Baseline, 4 weeks and 60 days
  The scale is scored by the patient's ability to complete specific tasks in daily life, including grooming, eating, bathing, dressing, stool control, urination control, toilet use, bed and chair transfer, walking on level ground, and going up and down stairs with 10 items.

CONTACTS AND LOCATIONS:
Overall Officials: RUJIE MA, Doctor, Study Director — The Third Affiliated hospital of Zhejiang Chinese Medical University
Locations (1):
- The Third Affiliated hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China